CLINICAL TRIAL: NCT06757556
Title: Effect of Consumption of Non-starchy Vegetables on Weight Status of Overweight and Obese University Population
Brief Title: Effect of Vegetables on Weight Status of University Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Qaisar Raza, Assistant Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Qaisar Raza
Record Dates: First submitted 2024-12-15; First posted 2025-01-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Obesity Control; Overweight and Obese Adults
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Interventional Randomized Controlled Trial.
Masking Description: There is no masking in this study as the participants are being informed whether they are in control or interventional group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre and post in-body assessment with no vegetable intake intervention. (No Intervention): Control group will consist of 20 participants and will be provided with no intervention. Pre assessment including in-body analysis of control group will be done in 1st week of study and post assessment will be done in 12th week of the study.
- Pre and post in-body assessment with vegetable intake intervention. (Experimental): Interventional group will consist of 20 participants. Pre assessment will be done in 1st week of study such as In-body analysis and intervention will be provided to these participants for 10 weeks and then post assessment will be done in 12th week after completion of intervention.
  2-3 servings (250g) of non-starchy vegetables, as recommended by WHO, will be provided to each participant for 10 weeks.
  Interventions: Other: Non-starchy vegetables will be provided to the participants as an intervention.

INTERVENTIONS:
Other: Non-starchy vegetables will be provided to the participants as an intervention. — Intervention will consist of provision of vegetables (based on WHO criteria of 2-3 servings) to overweight and obese adults fo weight loss purpose.
  Arms: Pre and post in-body assessment with vegetable intake intervention.

SUMMARY:
Obesity rates have more than doubled globally since 1990, with 2.5 billion overweight adults by 2022, and 890 million of them living with obesity (WHO, 2023). In Pakistan, approximately 30% of adults are overweight or obese, with 21% overweight and 9% obese. Non-communicable diseases now account for 58% of deaths in the country. WHO recommends daily consumption of non-starchy vegetables to aid weight loss and reduce BMI and fat mass, especially for overweight and obese individuals. This randomized controlled trial (RCT) will be conducted at the University of Veterinary and Animal Sciences (UVAS) in Lahore, Pakistan, targeting the university population, including students, teaching, and non-teaching staff with BMI ≥23 kg/m². A total of 40 participants will be recruited, with 20 assigned to the intervention group (receiving 2-3 cups of non-starchy vegetables daily) and 20 to the control group (receiving only dietary guidelines). Weight, BMI, and fat mass will be measured before and after the trial using an InBody 270. The data will be analyzed using SPSS version 25, with paired and independent t-tests to compare changes within and between groups. Multiple logistic regression will examine the relationship between vegetable consumption and changes in weight, BMI, and fat mass. This study aims to assess the impact of daily non-starchy vegetable intake on the weight, BMI, and fat mass of the overweight and obese university population.

DETAILED DESCRIPTION:
Obesity is an increasingly urgent public health challenge in both developed and developing countries. Since 1990, the global prevalence of adult obesity has more than doubled. By 2022, an alarming 2.5 billion adults (aged 18 years and older) were classified as overweight, with 890 million of them living with obesity (WHO, 2023). The World Health Organization (WHO) estimates that one in eight people worldwide now lives with obesity, which is linked to a variety of negative health outcomes, including increased risks for chronic diseases such as diabetes, hypertension, and cardiovascular conditions.

In Pakistan, the situation is equally concerning, with 30% of the adult population being either overweight or obese. More specifically, 21% of adults are classified as overweight, and 9% are considered obese. Non-communicable diseases (NCDs), such as heart disease, stroke, and diabetes, are now responsible for 58% of all deaths in the country. Overweight and obesity are particularly prevalent among young adults, whose sedentary lifestyle and poor dietary habits, including increased consumption of fast food and decreased vegetable intake, contribute significantly to weight gain. University students and staff in Pakistan are also heavily affected, with the prevalence of central obesity reaching 31.4% in males and 46% in females. In fact, 16% of Pakistani females and 30.5% of males have a BMI greater than or equal to 25 kg/m², as per local South Asian BMI cut-off points (Khan et al., 2016).

The WHO expert consultation in 2002 recommended lowering the BMI cut-off points for Asians to better address obesity-related public health concerns in the region, suggesting that a BMI of 23-27.5 kg/m² be classified as overweight, and a BMI of ≥27.5 kg/m² be categorized as obese (WHO, 2004). Given these statistics, there is a pressing need to identify effective, culturally appropriate interventions to combat obesity, particularly among university populations.

One promising intervention is increasing the intake of non-starchy vegetables, which are rich in nutrients and low in calories. WHO guidelines recommend daily consumption of non-starchy vegetables to aid weight management by improving overall diet quality, reducing fat mass, and lowering BMI. Research has shown that increasing vegetable consumption can help reduce body weight and fat mass, particularly in overweight and obese individuals.

This study aims to evaluate the effects of increasing daily non-starchy vegetable consumption on the weight, BMI, and fat mass of overweight and obese individuals in a university setting. A randomized controlled trial (RCT) will be conducted at the University of Veterinary and Animal Sciences (UVAS) in Lahore, Pakistan, involving students, teaching staff, and non-teaching staff who meet the inclusion criteria of a BMI ≥23 kg/m² based on South Asian cut-off points (Mahajan and Batra, 2018). A total of 40 participants will be randomly assigned to one of two groups: an intervention group and a control group, with 20 participants in each group.

The intervention group will receive 2-3 cups (approximately 250g) of WHO-recommended non-starchy vegetables daily for 10 weeks. These vegetables will include options like cucumbers, kale, cauliflower, spinach, cabbage, tomatoes, capsicum, broccoli, and lettuce, all of which have been shown to reduce body weight, BMI, and fat mass by influencing leptin levels (a hormone involved in regulating fat storage and hunger). The control group, on the other hand, will receive dietary guidelines on the recommended daily intake of non-starchy vegetables, but no vegetables will be provided.

Baseline assessments will be conducted during the first week of the study, where participants' weight, BMI, and fat mass will be measured using a weight scale and an InBody 270 body composition analyzer. Dietary counseling will also be provided at this stage, focusing on the benefits of non-starchy vegetables for weight management. From the second week onward, the intervention group will begin receiving their daily servings of vegetables, and the study will continue for 10 weeks.

At the conclusion of the 10-week intervention (week 12), post-assessment measurements will be taken for both the intervention and control groups. In addition to anthropometric measurements, participants in the intervention group will be asked to keep a food diary documenting their daily intake of non-starchy vegetables. This will help assess adherence to the intervention and track how participants incorporate the recommended vegetables into their daily diets.

The data collected will be analyzed using Statistical Package for Social Sciences (SPSS) version 25. Descriptive statistics will be used to present baseline measurements, while paired t-tests will compare changes within groups over the course of the study. Independent t-tests will assess differences between the control and intervention groups. Multiple logistic regression analysis will be employed to examine the relationship between non-starchy vegetable consumption and changes in weight, BMI, and fat mass, controlling for confounding variables such as other dietary factors.

This study seeks to provide valuable insights into the effectiveness of increasing non-starchy vegetable intake in reducing weight, BMI, and fat mass among overweight and obese university populations in Pakistan. The findings could have important implications for public health initiatives aimed at addressing obesity and improving diet quality in university settings, contributing to broader efforts to combat the obesity epidemic in South Asia.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese individuals with BMI 23kg/m^2
* Population of UVAS (students, teaching and non-teaching staff)

Exclusion criteria:

* Normal weight and underweight individuals with BMI <23kg/m^2
* Non-UVAS (University of Veterinary and Animal Sciences) population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-09-08 (Estimated)

PRIMARY OUTCOMES:
Weight status (BMI) | 12 weeks
  Intervention consists of provision of vegetables based on WHO criteria of 2-3 servings (250g) for weight loss purposes. the Investigator will calculate the body mass index of participants which is the general indicator of weight status.

SECONDARY OUTCOMES:
Fat mass (Percent body fat) | 12 weeks
  The investigator will check the percentage of body fat in relation to the total body weight of the participants. Percentage body fat is the measure of amount of fat in your body compared to your lean body mass (muscle, bone, water etc).

CONTACTS AND LOCATIONS:
Overall Officials: Qaisar Raza, PhD, Principal Investigator — UVAS Lahore
Locations (1):
- Qaisar Raza, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be shared in the form of a thesis to be submitted to the university (UVAS, Lahore, Pakistan) and in the form of research papers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD information will be shared by June 2025 and will be available indefinitely.
Access Criteria: IPD information will be available for researchers and general public through electronic and print sources.

REFERENCES:
- See also: The information will be shared in the form of thesis on this website — https://uvas.edu.pk/